CLINICAL TRIAL: NCT03784352
Title: Virtual Reality in Reducing Pain and Anxiety in Pediatric Orthopaedics, a Pilot Randomized Controlled Trial
Brief Title: Virtual Reality Pediatric Orthopaedic Outpatient Procedures
Acronym: VPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Children's Hospital (Other)
Responsible Party: Principal Investigator, Bejaan Jivraj, Research Student, British Columbia Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-03184
Record Dates: First submitted 2018-12-13; First posted 2018-12-21 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) (Experimental): The intervention will consist of standard of care (SOC) in addition to the use of virtual reality. SOC consists of the technician/care provider explaining the procedure while using speech to be comforting and supportive in addition to parent/guardians being allowed to console and distract their child during the procedure and interacting with other distractions techniques that may be available (ie. ipad, or mobile device) Patients assigned to the VR group will interact with VR through mobile-based VR googles.
  Interventions: Device: Virtual Reality
- No Virtual Reality (VR) (No Intervention): This arm will receive regular standard of care (SOC), the same that would be received if they were not enrolled in the study. SOC will include the technician/care provider explaining the procedure while using speech to be comforting and supportive in addition to parent/guardians being allowed to console and distract their child during the procedure and interacting with other distractions techniques that may be available (ie. ipad, or mobile device)

INTERVENTIONS:
Device: Virtual Reality — A calming virtual reality game will be played
  Arms: Virtual Reality (VR)

SUMMARY:
The main objective of the study is to evaluate the use of Virtual Reality (VR) in managing pain and anxiety levels during common pediatric orthopaedic outpatient procedures which include: cast application, cast removal, hardware removal (ie. pins and screws), and botox injections.

DETAILED DESCRIPTION:
Immediately following recruitment, demographic data and diseased related information (ie. location of cast/hardware, reason for cast/hardware placement and location and reason for botox injection) will be collected through self and/or guardian report. All data will be collected using REDCap (research electronic data capture). Using a parallel group design, patients will then be stratified by age (4-7, 8-12 and 13-18 years), gender, and procedure classifications (hardware or cast or staple or suture removal or cast application or botox injection) site of hardware or cast or staple or suture or botox injection), and reason for the procedure (trauma vs a preexisting orthopaedic condition). After randomization by the REDCap system, patients are taken into the procedure room where a questionnaire (Short STAI) is completed by the patient to collect pre-procedural state anxiety measurements. Following this, patients in the control group will receive standard of care (SOC) which allows for the technician and/or accompanying guardian to try and distract and or console the patient as they normally would. The patients in the intervention group will receive SOC with Virtual Reality (VR) interaction a few minutes before, during and following the procedure (around 5-10minutes total). During the procedure the researcher will complete an observational survey (CEMS) to assess procedural state anxiety. Upon completion, both groups will then be asked to complete a survey (Short STAI) to collect post-procedural anxiety levels and an additional survey (Wong Baker Scale) to retrospectively collect pain levels from during the procedure and their current pain levels post procedure while parent/guardians and cast technician will be asked to complete their respective satisfaction questionnaires. Following this, the child will be asked if they experienced any nausea at any point during the procedure, if they did, they will be asked to complete the BARF questionnaire to measure the amount of nausea experienced. Following completion of questionnaires, patients who were in the control group are invited to interact with the VR simulation for a total of 5 minutes. This was chosen to incentivize recruitment for the study.

SOC will consist of the technician/care provider explaining the procedure while using speech to be comforting and supportive in addition to parent/guardians being allowed to console and distract their child during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* child must be between the ages of 4 and 18 years
* the parent/guardians and child are both able to speak and read English or have a translator be present for them

Exclusion Criteria:

* symptoms of respiratory or gastrointestinal infection
* visual, auditory, cognitive impairment or developmental delay
* history of seizures or epilepsy

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Wong Baker Scale (WBS) for Procedural Pain | Immediately post procedure
  The WBS is a self-reported outcome measure that asks patients to rate their pain severity by circling the face that best describes the pain on a horizontally positioned VAS with marked end points of "no pain" and "worst possible pain". There are six possible faces with "no pain" representing a score of 0 and "worst pain" representing a score of 10
Anxiety (state anxiety intraprocedure) | Intraprocedure
  Intraprocedural state anxiety will be measured using the The Children's Emotional Manifestation Scale (CEMS) which consists of five categories that include:
  Facial expression, vocalization, activity, interaction and level of cooperation. A score is obtained by reviewing five descriptions in each category and selecting the number that most clearly represents the observed behavior. Each category is given a score from 1 to 5 for a total score of 5-25. A higher score corresponds to a more distressed child.

SECONDARY OUTCOMES:
Procedural Time | Intraprocedure
  Measured with a stopwatch: Start of the procedure defined as the moment the patient completes the first short SAIS, which is shortly upon entering the procedural room. End of the procedure is marked as follows: complete removal of cast (for cast removal), removal of last staple or hardware (staple and hardware removal), removal of needle from final injection site (botox injection)
Baxter Retching Faces (BARF) Scale for Nausea | Immediately post procedure
  Patients will use the pictorial Baxter Retching Faces Scale (BARF) to measure nausea severity. It is a scale of 0-10 with 6 faces, with the first representing no nausea to the last as experiencing vomiting. This scale has been shown to have construct, content and convergent validity in measuring nausea in children. After the patients have completed the post procedure short SAIS the patients will be asked if they had experienced any feelings of nausea at any point during the procedure. If they answer yes, then they will be asked to rate the nausea using the BARF scale.
State Anxiety Preprocedure | Immediately pre-procedure
  State Anxiety will be measured prior to start of procedure using the Short SAIS (state anxiety inventory scale) which is a shortened version of the Spielberger State Trait Anxiety Inventory (STAI) Scale will be used to collect data on state anxiety. State anxiety refers to the anxiety levels at a particular moment in time. This is in contrast to trait anxiety which is a measure of the tendency of an individual to experience anxiety across different situations. The short SAIS is a six item questionnaire with four possible responses for each item. The total score ranges from 6-24 points, with 6 points indicating no anxiety and 24 points indicating the highest level of anxiety. The total time to complete the questionnaire is approximately five minutes.
State Anxiety Postprocedure | Immediately post procedure
  State Anxiety will also be measured immediately after completion of the procedure using the Short SAIS (state anxiety inventory scale) which is a shortened version of the Spielberger State Trait Anxiety Inventory (STAI) Scale will be used to collect data on state anxiety. State anxiety refers to the anxiety levels at a particular moment in time. This is in contrast to trait anxiety which is a measure of the tendency of an individual to experience anxiety across different situations. The short SAIS is a six item questionnaire with four possible responses for each item. The total score ranges from 6-24 points, with 6 points indicating no anxiety and 24 points indicating the highest level of anxiety. The total time to complete the questionnaire is approximately five minutes.
Trait Anxiety | Preprocedure while in the waiting area
  The Penn State Worry Questionnaire for Children (PSWQ-C) is a screening tool for assessing generalized anxiety in children aged 7-17 years. It consists of a 14 item self-reported questionnaire. Respondents indicate how often each item applies to them, choosing from the following responses: "never", "sometimes", "often", and "always", with points ranging from 0 to 3 for each item. The total score ranges from 0 to 42, with higher scores indicating a greater tendency to worry. The total time to complete the questionnaire is approximately five minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, MBBS, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No